CLINICAL TRIAL: NCT06318533
Title: An Exploratory Clinical Study of the Safety and Efficacy of CD19 Chimeric Antigen Receptor NK Cell Injections for the Treatment of Relapsed/Refractory B-cell Related Autoimmune Diseases
Brief Title: A Clinical Study of CD19 CAR NK Cells for the Treatment of Relapsed/Refractory B-cell Related Autoimmune Diseases
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: YANRU WANG (Other)
Collaborators: Rui Therapeutics Co., Ltd (Industry)
Responsible Party: Sponsor-Investigator, YANRU WANG, Director, Department of Rheumatology and Immunology, Affiliated Hospital of Jiangsu University
Organization: Affiliated Hospital of Jiangsu University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-11-01
Record Dates: First submitted 2024-03-12; First posted 2024-03-19 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Autoimmune Diseases
MeSH Terms: conditions — Autoimmune Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-CD19 CAR NK cells (Experimental)
  Interventions: Drug: anti-CD19 CAR NK cells

INTERVENTIONS:
Drug: anti-CD19 CAR NK cells — Patients will receive Fludarabine (30mg/m2 per day) and Cyclophosphamide (300mg/m2 per day) on day -5, -4, and -3, followed by Anti-CD19 CAR NK cells infusion.

SUMMARY:
A single arm, open-label pilot study is designed to determine the safety and effectiveness of anti-CD19 CAR NK cells (KN5501) in patients with relapsed/refractory B-cell related autoimmune diseases.15 patients are planned to be enrolled in the dose-escalation trial (6×10^9 cells, 9×10^9 cells). The primary objective of the study is to evaluation of the safety and feasibility of KN5501 for the treatment of relapsed/refractory B-cell related autoimmune diseases. The secondary objective is to evaluate the effectiveness of KN5501 for the treatment of relapsed/refractory B-cell related autoimmune diseases. The exploratory objective is to evaluate expansion, persistence and ability to deplete CD19 positive B cells of KN5501 in patients with relapsed/refractory B-cell related autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects voluntarily participate in this clinical study and sign the Informed Consent Form (ICF) and are willing to follow and be able to complete all trial procedures
2. Subjects disease status of enrolment: not complete response (CR) after standard treatment; moderately to severely active autoimmune diseases
3. Age: ≥ 18 years old and ≤ 70 years old, male or female
4. Subjects with estimated survival > 12 weeks
5. Adequate organs function: Serum creatinine clearance meets relevant age/sex criteria,aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 times the upper limit of normal (ULN)
6. ECOG performance ≤ 2
7. Left ventricular ejection fraction (LVEF) ≥ 45%
8. Subjects have been treated with OCS in combination with an immunosuppressive or biologic agent for at least 2 weeks prior to enrollment

Exclusion Criteria:

1. Subjects with known severe allergic reactions, hypersensitivity, contraindication to any medications during the trial (cyclophosphamide, fludarabine, tozumabs), or subjects with a history of severe allergic reactions
2. Subjects with one of the following genetic syndromes: Fanconi syndrome, Kostmann syndrome, Shwachman syndrome or any of the known bone marrow failure syndromes
3. Subjects with active or uncontrolled infections requiring parenteral antimicrobials; evidence of severe active viral or bacterial infections or uncontrolled systemic fungal infections
4. Subjects with grade III or IV heart failure (NYHA classification)
5. History of epilepsy or other central nervous system (CNS) diseases
6. History of other primary malignant tumors except: cured non-melanoma skin cancer or primary cervical cancer; subjects with inactive tumors
7. Subjects with more pronounced bleeding tendencies, such as gastrointestinal bleeding, coagulation disorders, and hypersplenism
8. Subjects were treated with systemic corticosteroids concomitantly within 2 weeks prior to treatment
9. Subjects with unstable angina, symptomatic congestive heart failure or myocardial infarction within the last 6 months
10. Females who are pregnant, lactating, or planning a pregnancy within six months
11. Subjects who have received other clinical trial treatment within 3 months
12. Any situation judged by the investigators that may increase the risk of the subjects or interfere with the clinical trial outcome

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2026-03-13 (Estimated); Study Completion 2027-03-13 (Estimated)

PRIMARY OUTCOMES:
Incidence of Dose Limiting Toxicity (DLTs) | within 4 weeks after infusion; 12, 24, 36 and 52 weeks after infusion
  To characterize the safety of anti-CD19 CAR NK Cells for moderate to severe autoimmune diseases.
Treatment Emergent Adverse Events（TEAEs） | within 4 weeks after infusion; 12, 24, 36 and 52 weeks after infusion
  To characterize the safety of anti-CD19 CAR NK Cells for moderate to severe autoimmune diseases

SECONDARY OUTCOMES:
Disease control rate of subjects | 4, 12, 24, and 52 weeks after infusion
  To characterize the efficacy of anti-CD19 CAR NK Cells for moderate to severe autoimmune diseases. Disease control is assessed according to SLEDAl 2K. Disease control rate is defined as proportion of patients with SRI-4 response: including SLEDAI 2K ≥ 4-Point improvement
Remission rate of subjects | 4, 12, 24, and 52 weeks after infusion
  To characterize the efficacy of anti-CD19 CAR NK Cells for moderate to severe autoimmune diseases. Remission is assessed according to SLEDAl 2K. Remission rate is defined as proportion of patients with SLEDAl 2K score= 0

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - Jiangsu University Affiliated Hospital, Zhenjiang, Jiangsu

IPD SHARING:
Plan to Share IPD: No